CLINICAL TRIAL: NCT00449969
Title: Quality of Out-of-hospital Cardiopulmonary Resuscitation (CPR) With Real Time Automated Feedback: a Prospective Randomized Study
Brief Title: Out-of-hospital Cardiopulmonary Resuscitation and AED Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Thomas P. Weber, principle investigator, Department of Anesthesiology and Intensive Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-AnIt-07
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Cardiac Arrest; Resuscitation
Keywords: AED (automated external defibrillation); feedback; out of hospital resuscitation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Extended feedback (Experimental)
  Interventions: Device: Zoll AED pro
- 2. Limited feedback (Active Comparator)
  Interventions: Device: Zoll AED pro

INTERVENTIONS:
Device: Zoll AED pro — Arm one (Extended feedback) offers full feedback guidance during CPR
  Arms: 1. Extended feedback
Device: Zoll AED pro — In arm two (limited feedback) feedback is modified lacking several elements of feedback
  Arms: 2. Limited feedback

SUMMARY:
The purpose of this study is to determine whether an online automatic feedback improved CPR quality (No-flow time, compression depth, short-term survival and one year follow up) in this prospective randomised study of out-of-hospital cardiac arrest

ELIGIBILITY:
Inclusion Criteria:

* cardiac arrest

Exclusion Criteria:

* age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
ratio of patients with spontaneous circulation | admission to the hospital

SECONDARY OUTCOMES:
length of hospital stay | hospital discharge
neurological status | hospital discharge
neurological status | one year after resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Weber, MD, Study Chair — Department of Anesthesiology and Intensive Care, University Hospital Muenster
Locations (1):
- Department of Anesthesiology and Intensive Care, University Hospital Muenster, Münster, Germany

REFERENCES:
- [Result] Lukas RP, Sengelhoff C, Dopker S, Harding U, Mertens P, Osada N, Van Aken H, Weber TP, Bohn A. [Chest compression quality : Can feedback technology help?]. Anaesthesist. 2010 Feb;59(2):135-9. doi: 10.1007/s00101-009-1671-4. German. PMID 20151103
- [Result] Bohn A, Weber TP, Wecker S, Harding U, Osada N, Van Aken H, Lukas RP. The addition of voice prompts to audiovisual feedback and debriefing does not modify CPR quality or outcomes in out of hospital cardiac arrest--a prospective, randomized trial. Resuscitation. 2011 Mar;82(3):257-62. doi: 10.1016/j.resuscitation.2010.11.006. Epub 2010 Dec 13. PMID 21146279